CLINICAL TRIAL: NCT05873881
Title: COLchicine and Thiamine in Heart Failure Due to Ischemic Heart Disease
Acronym: COLT-HF
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Population Health Research Institute (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: PHRI.COLT-HF
Record Dates: First submitted 2023-05-15; First posted 2023-05-24 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Colchicine; Thiamine

STUDY DESIGN:
Intervention Model Description: Factorial 1: Colchicine 0.5 mg daily or placebo Factorial 2: Thiamine 300mg daily or no thiamine
Who Masked: Participant, Outcomes Assessor
Masking Description: Factorial 1: Placebo controlled. Factorial 2: Prospective Randomized Open Blinded End-point (PROBE) design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Colchicine versus placebo (Placebo Comparator): Randomization to colchicine or placebo
  Interventions: Drug: Colchicine 0.5 MG; Drug: Colchicine placebo
- Thiamine versus no thiamine (Experimental): Randomization to thiamine or to no thiamine in a PROBE design
  Interventions: Drug: Thiamine Mononitrate 300 mg

INTERVENTIONS:
Drug: Colchicine 0.5 MG — Oral colchicine 0.5 mg daily
  Arms: Colchicine versus placebo
Drug: Colchicine placebo — Placebo colchicine daily
  Arms: Colchicine versus placebo
Drug: Thiamine Mononitrate 300 mg — Thiamine Mononitrate 300 mg daily
  Arms: Thiamine versus no thiamine

SUMMARY:
The goal of this 2x2 factorial clinical trial is to test the efficacy of i) colchicine, and ii) thiamine in heart failure (HF) secondary to ischemic heart disease. The main questions it aims to answer are:

* Does colchicine reduce the risk of cardiovascular (CV) death, a HF event, or an ischemic CV event
* Does thiamine reduce the risk of cardiovascular (CV) death, or a HF event

Participants will undergo the following procedures:

* Run-in: All participants will receive colchicine 0.5 mg daily to assess drug tolerance over a 3-4 week period.
* Randomization: If colchicine is tolerated during run-in, eligible participants will be randomized in a 2x2 factorial design to receive i) colchicine 0.5mg daily or placebo, and ii) thiamine 300mg daily or no thiamine.
* Follow-up: Clinical outcomes, side effects, adverse events, and drug adherence will be captured during follow-up

ELIGIBILITY:
Inclusion Criteria:

1. Age >/= 45 years
2. Documented ischemic HF as the etiology of HF, which includes:

   1. a prior history of CAD (defined as a history of myocardial infarction, coronary artery bypass graft surgery, percutaneous coronary intervention, or non-invasive or invasive cardiac testing consistent with a diagnosis of CAD), and
   2. determination of CAD to be the cause primary cause of HF based on local investigator assessment
3. New York Heart Association (NYHA) class II-IV symptoms
4. Documented LVEF </= 45% within 1 year prior to enrollment
5. Optimization of HF treatment based on local practice.
6. Ambulatory HF patients or stable hospitalized patients with HF will both be eligible for enrollment in the trial. For hospitalized patients, enrollment will require i) evidence of clinical stability from HF defined as no use of an inotropic agent or intravenous diuretic agent in the prior 24, and ii) expected discharge from hospital in the next 72 hours.

Exclusion Criteria:

1. Female who is pregnant, breast-feeding, or of childbearing potential and not using an effective form of birth control*
2. Regular or required use colchicine or thiamine for other clinical indications.**
3. History of allergic reaction to colchicine or to thiamine; or current or planned use of cyclosporine, verapamil, diltiazem, azole antifungal, macrolide antibiotic (except azithromycin), or HIV protease inhibitor
4. Use of a ventricular assist device or prior heart transplant
5. Coronary revascularization (coronary artery bypass graft surgery or percutaneous coronary intervention) within the 4 weeks prior to enrollment, or planned within the next 4 weeks.
6. Severe valvular disease
7. Chronic and severe renal dysfunction defined as eGFR < 15 mL/min/1.73m2 based on local laboratory measurement done within 6 months prior to run-in***
8. History of liver cirrhosis
9. Active malignancy (excluding basal cell or treated squamous cell carcinoma of the skin) requiring treatment and with a life-expectancy of < 2 years.
10. Concurrent use of other experimental pharmacologic agents -

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Colchicine arm: Time to first occurrence of a CV death, a HF event, MI, stroke, or arterial revascularization | 3.5 years
Thiamine arm: Time to first occurrence of a CV death, or a HF event | 3.5 years

SECONDARY OUTCOMES:
Time to death | 3.5 years
Time to first hospitalization | 3.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Philip G Joseph, M.D., Principal Investigator — Population Health Research Institute
Locations (1):
- Hamilton Health Sciences Corporation, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No